CLINICAL TRIAL: NCT01313533
Title: Biologically Modified Saphenous Vein Transplants for Improved CABG Outcomes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Luke's Hospital, Chesterfield, Missouri (Other)
Responsible Party: Principal Investigator, Ron Fiehler, Biologically Modified Saphenous Vein Transplants for Improved CABG Outcomes, St. Luke's Hospital, Chesterfield, Missouri
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R9-LRS-CS-01
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Atherosclerosis
Keywords: Atherosclerosis of Autologous Vein Bypass Graft
MeSH Terms: conditions — Atherosclerosis | interventions — polyarginine; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactated Ringers Solution with Arginine (Active Comparator): 100 ml of LRS with arginine
  Interventions: Drug: Polyarginine
- Lactated Ringers Solution (Placebo Comparator): Lactated ringers solution
  Interventions: Drug: Vein soak treated with Lactated Ringers Solution

INTERVENTIONS:
Drug: Polyarginine — Vein soak treated with polyarginine
  Arms: Lactated Ringers Solution with Arginine
Drug: Vein soak treated with Lactated Ringers Solution — Vein soak
  Arms: Lactated Ringers Solution

SUMMARY:
The purpose of this study is to study the effects of polyarginine treated vein grafts on graft patency for patients undergoing coronary artery bypass surgery.

DETAILED DESCRIPTION:
Double blind study with Lactated Ringers Solution and Lactated Ringers Solution with Arginine soaked for 10 minutes prior to grafting on the coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 25-95 years of age and able to give informed consent
2. Use of an approved statin and anti-platelet medication for at least 24 months.
3. Agreeable to Cardiovascular imaging at 12 months post-coronary artery bypass graft (CABG).
4. First time coronary artery bypass surgery,redo coronary artery bypass surgery and combined valve repair/replacement surgery and coronary artery bypass graft surgery are eligible to participate in study.

Exclusion Criteria:

1. Acute traumatic injury, vasculitis or planned concurrent ventricular surgical restoration, automatic implantable cardioverter defibrillators (AICD) placement or valvular surgery.
2. Hypercoaguable state.
3. Comorbid illness making 2 year survival unlikely.
4. Participation in another interventional investigative study of a cardiovascular drug or device within 30 days prior to CABG. May participate concurrently in other studies where the intervention/observation will not hinder execution of this study.
5. Patients with any medical condition that, in the investigator's judgment, makes the patient ineligible or places the patient at undue risk (e.g. conditions that preclude standard invasive follow up procedures such as angiography, i.e. renal failure, bleeding diathesis or peripheral vascular disease preventing catheterization via the groin).
6. Subject has clinical evidence of infection that the Investigator deems significant to the completion of the procedure or that could compromise the subject's safety.
7. Any patient was has undergone more than 20 computerized tomography (CAT) scans.
8. Any patient who is pregnant.

Ages: 25 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-12 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
To study the effects of arginine on saphenous vein graft patency rates | 12 months post operation
  To study the effects of arginine on saphenous vein graft patency rates

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Leidenfrost, MD, Principal Investigator — St. Luke's Hospital
Locations (1):
- St. Luke's Hospital, Chesterfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided